CLINICAL TRIAL: NCT03938428
Title: The Patient Experience of a Paramedic-Pharmacist Referral Pathway for Clinical Medication Reviews
Acronym: PEPPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yorkshire Ambulance Service NHS Trust (Other Government)
Collaborators: NIHR Yorkshire and Humber Patient Safety Translational Research Centre (Unknown)
Responsible Party: Sponsor
Other Study IDs: YASRD114; 263976 (Other: IRAS)
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Pharmaceutical Preparations; Accidental Fall; Allied Health Personnel
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Patients who are eligible for this study will have been previously identified as part of the PREFACES project. The pharmacist who has conducted the clinical medication review will obtain verbal permission from the patient to be contacted by the research study team. This will be documented on the referral outcome document that is returned to the YAS clinical team. A member of YAS clinical staff from the PREFACES project will forward the name and residential address of patients who have agreed to be contacted to the research paramedic for this study. A covering letter, participant information sheet, questionnaire and consent form, will be posted to potential participants. A stamped addressed envelope will be included to enable return of the completed booklet at no costs to participants.

SUMMARY:
This study seeks to understand how patients feel about their medicines before and after receiving a clinical medication review.

DETAILED DESCRIPTION:
Falls in people aged 65 years and over are a common reason for calling the emergency ambulance service. Falls can be serious, with about 1 in 20 people having to be taken to hospital because they have been injured. Thankfully, in more than 4 out of 10 cases, people are not seriously injured and can be left at home. However, it is important that the reason for the fall is found and future falls are prevented where possible.

Yorkshire Ambulance Service can already make a referral to another local service to get specialist practical help for falls prevention when people are left at home after a fall. Research has shown that the safe use of medicines can prevent future falls, but that did not form. Now a new service has been set up for Yorkshire Ambulance Service to refer patients to the Leeds GP Confederation. A pharmacist working in the patients GP surgery will undertake a review of the patient's use of their medicines.

We would like to find out about how patients feel about using their medicines before and after the medicines review by a pharmacist. We would also like to know how they feel about the medicines review itself, to help decide whether this scheme should continue or be expanded to other areas. To do this, we are going to send a questionnaire to patients who receive a medicines review. The questionnaire will be sent by post, take about 10 minutes to fill out and include a stamped addressed envelope so people who take part will not have to pay for postage.

ELIGIBILITY:
Inclusion Criteria:

* Received a pharmacist-led clinical medication review following a falls referral made by a paramedic from Yorkshire Ambulance
* Registered with a GP in the Leeds area
* Has capacity to consent to take part in the study

Exclusion Criteria:

* Did not receive a pharmacist-led clinical medication review after a Yorkshire Ambulance Service paramedic made a falls referral
* Not registered with a GP in the Leeds area
* Does not have capacity to consent to take part in the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted from a single site (Yorkshire Ambulance Service NHS Trust). YAS staff make around 70-100 falls referral pathways a month in the Leeds area, and after exclusions relating to the PREFACS projects, it is anticipated that around 55 patients per month will be eligible to receive a pharmacist-led clinical medication review and will therefore be eligible for this study, up to a maximum of 550 patients.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who express a change in emotion relating to how they feel about their medicines, following a pharmacist-led clinical medication review. | 1 month

SECONDARY OUTCOMES:
Patient expressed emotion | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Yorkshire Ambulance Service NHS Trust, Wakefield, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No